CLINICAL TRIAL: NCT00099515
Title: Standard Training Versus Intensive Training for HIIP Delivery System Usage in Insulin-Naïve Patients With Type 2 Diabetes Mellitus
Brief Title: Comparing Intensive and Standard Training for Human Insulin Inhalation Powder (HIIP)
Acronym: IDAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Alkermes, Inc. (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9523; H7U-MC-IDAP
Record Dates: First submitted 2004-12-15; First posted 2004-12-16 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: LY041001 (HIIP)
- B (Experimental)
  Interventions: Drug: LY041001 (HIIP)

INTERVENTIONS:
Drug: LY041001 (HIIP) — Inhalation, capsule, TID 3 times per day min 6 IU max 60 IU
  Arms: A
Drug: LY041001 (HIIP) — Inhalation, Capsule, TID 3 times per day min 6 IU max 60 IU
  Arms: B

SUMMARY:
The purpose of this study is to compare intensive and standard training for human insulin inhalation powder in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 12 months
* Age 18 or older.
* Taking at least 1 oral antihyperglycemic medication.
* Have an HbA1C between 7.5 and 12.
* Be a nonsmoker

Exclusion Criteria:

* Body Mass Index (BMI) greater than 40.
* Have frequent episodes of severe hypoglycemia.
* Have advanced autonomic neuropathy.
* Have history of asthma.
* Have chronic obstructive pulmonary disease (COPD).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2004-11; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Hypothesis that std training for HIIP system is noninferior to intensive training by 1.2 mmol/L with respect to overall 2-hr postprandial glucose excursion of (SMBG) in type 2 diabetes patients that have been on preprandial trmt with HIIP | 4 weeks

SECONDARY OUTCOMES:
Assess the suitability of the HIIP delivery system for type 2 diabetes patients | 4 weeks
Compare the SMBG profiles of preprandial HIIP administration with standard training and with intensive training Assess patient compliance with the HIIP delivery system Directions for Use (DFU) provided by the Sponsor with and without intensive training | 4 weeks
Compare the test meal blood glucose profiles of preprandial HIIP administration with standard training and with intensive training | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clearwater, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buffalo, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Hyde Park, New York
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sante Fe, Rosario, Argentina
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norway, Portugal
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., George, South Africa

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com